CLINICAL TRIAL: NCT06485505
Title: Efficacy of Low Dose Isotretinoin Versus Excimer Light as an Adjuvant for Itraconazole in Treatment of Onychomycosis: a Randomized Controlled Trial.
Brief Title: Isotretinoin Versus Excimer Light an Adjuvant in Treating Onychomycosis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mona El Radi Kamal Mohamed Emam, Principle Investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Onychomycosis
Record Dates: First submitted 2024-05-30; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — Isotretinoin; Itraconazole

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Itraconazole (Active Comparator): all patients will be prescribed Itraconazole in the dose of 200mg twice daily for 1 week per month, for 3 consecutive months after screening of complete blood count, liver, and renal function tests. patients were advised to record any side effects
  Interventions: Drug: Itraconazole 200 mg
- Itraconazole + Low dose Isotretinoin (Experimental): patients will be given low dose of isotretinoin as an adjuvant to itraconazole in the same previously mentioned protocol. Treatment protocol consists of low dose isotretinoin (20mg, every other day for pediatrics) for a 3- month course. After completion of the course, treating dose of isotretinoin was maintained for 4-6 weeks to prevent recurrence, and to improve healing. During treatment, an infrequent application of the previous therapies was permitted.
  Interventions: Drug: ISOtretinoin 10 MG
- Itraconazole +Excimer light (Experimental): will be treated with excimer light as an adjuvant to itraconazole in the same previously mentioned protocol. Nails will be treated with XeCl2 excimer light (Eximal Elite Device).
  Interventions: Device: excimer light

INTERVENTIONS:
Drug: ISOtretinoin 10 MG — Low dose isotretinoin as an adjuvant for itraconazole in treating onychomycosis
  Arms: Itraconazole + Low dose Isotretinoin
Device: excimer light — excimer light as an adjuvant for itraconazole in treating onychomycosis
  Arms: Itraconazole +Excimer light
Drug: Itraconazole 200 mg — Itraconazole alone
  Arms: Itraconazole

SUMMARY:
3 groups of patients with onychomycosis will be recruited. Group A will receive itraconazole alone. Group B will receive itraconazole + low dose isotretinoin and group C will be treated with itraconazole + excimer light sessions.

DETAILED DESCRIPTION:
The sample size will be calculated by a statistician based upon the rate of onychomycosis cases attending at the outpatient clinical. 3 equal groups of patients will be included. inclusion criteria include: -definite diagnosis of dermatophyte onychomycosis using KOH examination and a fungal culture - a washout period of at least 1 month of any previous therapy -age> 16 years Exclusion criteria include: -pregnancy and lactation -Any active infection or inflammation in or around the nails other than onychomycosis -patients with liver diseases, heart disease and diabetes

Steps of performance and techniques used:

1. Complete history taking.
2. Detailed local examination:

Local examination will be done for the nail to detect swelling, induration, erythema around the nail, local pain and presence of pus during the sessions.

Patients with proven onychomycosis clinically, dermoscopically and through culture will be included in the study.

The included patients will sign an informed written consent before the beginning of the study, and the study will be done under the approval of the ethical committee for postgraduate studies and research of faculty of Medicine, Zagazig University.

Onychomycosis severity index (OSI) will be used for grading of onychomycosis severity where 0=no onychomycosis,1-5= mild onychomycosis,6- 15=moderate onychomycosis, and 16-35=severe onychomycosis.

The patients will be divided into 3 equal groups:

GROUP 1: (itraconazole group); all patients will be prescribed Itraconazole in the dose of 200mg twice daily for 1 week per month, for 3 consecutive months after screening of complete blood count, liver, and renal function tests. patients were advised to record any side effects.

GROUP 2 : will be given low dose of isotretinoin as an adjuvant to itraconazole in the same previously mentioned protocol.

Treatment protocol consists of low dose isotretinoin 20mg, every other day for a 3- month course. After completion of the course, treating dose of isotretinoin will be maintained for 4-6 weeks to prevent recurrence, and to improve healing. During treatment, an infrequent application of the previous therapies will be permitted.

GROUP 3: will be treated with excimer light as an adjuvant to itraconazole in the same previously mentioned protocol. Nails will be treated with XeCl2 excimer light (Eximal Elite Device).

ELIGIBILITY:
Inclusion Criteria:

* patients with onychomycosis

Exclusion Criteria:

* pregnant and lactating females patients on statin therapy or photosensitizing drugs patients with liver disease, heart disease and diabetes milletus.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Clinical improvement | 6 month frame: clinical assessment will be done at first presentation of the patients, monthly during the treatment course, at the last visit and 3 month after stoppage of treatment at the follow up visit in a total span of 6 months
  using onychomycosis severity index at baseline, last session and follow up vistis
Culture | 6 month frame: Fungal culture will be done at first presentation of the patients, at the last visit and 3 month after stoppage of treatment at the follow up visit in a total span of 6 months
  Fungal culture to detect fungal cause and presence after treatment

IPD SHARING:
Plan to Share IPD: No